CLINICAL TRIAL: NCT05618782
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Trial of the Efficacy and Safety of LEVI-04 in Patients With Osteoarthritis of the Knee
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of LEVI-04 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Levicept (Industry)
Collaborators: Nordic Bioscience Clinical Development (NBCD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEVI-04-21-02
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pain; Osteo Arthritis Knee; Knee Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Osteoarthritis; Knee; Levi-04
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial of multiple doses and multiple administrations of LEVI-04 for the treatment of pain due to osteoarthritis of the knee. The study consists of a Screening Period (including a Diary Run- In/analgesic wash-out Period), Randomization, Post-Randomization Period, and a Follow-up Period. Up to 624 participants will be enrolled and randomized to one of four Treatment Arms at the ratio 1:1:1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double- Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.3 mg/kg LEVI-04 (Active Comparator): Intravenous infusion of 0.3 mg/kg LEVI-04
  Interventions: Drug: LEVI-04
- 1.0 mg/kg LEVI-04 (Active Comparator): Intravenous infusion of 1.0 mg/kg LEVI-04
  Interventions: Drug: LEVI-04
- 2.0 mg/kg LEVI-04 (Active Comparator): Intravenous infusion of 2.0 mg/kg LEVI-04
  Interventions: Drug: LEVI-04
- Placebo (Placebo Comparator): Intravenous infusion of saline vehicle as placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LEVI-04 — LEVI-04, a fully human chimeric fusion protein that combines the Fc fragment of human immunoglobulin G1 with the p75 neurotrophin receptor (p75 NTR), for the treatment of chronic pain.
  Arms: 0.3 mg/kg LEVI-04; 1.0 mg/kg LEVI-04; 2.0 mg/kg LEVI-04
Other: Placebo — Saline vehicle
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, double-blind, placebo-controlled trial of multiple doses and multiple administrations of LEVI-04 for the treatment of pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
The study consists of a Screening Period (including a Diary Run- In/analgesic wash-out Period), Randomization, Post-Randomization Period, and a Follow-up Period. Up to 624 participants will be enrolled and randomized to one of four Treatment Arms at the ratio 1:1:1:1

The overall objective of this study is to evaluate the efficacy and safety of LEVI-04 compared to placebo in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent form (ICF).
2. Male or female participants between ≥40 and ≤80 years of age.
3. BMI ≤40 kg/m2.
4. The ability to utilize the eDiary device provided by study sites.
5. History of knee pain on most days for at least 3 months prior to Screening
6. Confirmation of OA of the knee

   1. Radiographs of both knees with a Posterior-Anterior, Fixed-flexion view taken during the Screening Period.
   2. American College of Rheumatology (ACR) clinical and radiographic diagnostic criteria.
7. Evidence of knee OA with a KL grade ≥2, determined through central reading.
8. Target Knee must have a score of ≥20 out of 50 on the WOMAC pain subscale during Screening and at Randomization
9. The Baseline (NRS) Pain score will be derived from the last seven days of the Diary Run-In Period and must meet following criteria:

   1. Completion of Average Daily (NRS) Pain score on at least 6 of the 7 days.
   2. Mean Average Daily (NRS) Pain score must be ≥4.0 and ≤9.0
   3. Mean Average Daily (NRS) Pain variability must be ≤1.5
10. If female, not of childbearing potential defined as post-menopausal for at least 1 year, or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practicing an agreed upon highly effective method of birth control throughout the study period.
11. If male and sexually active with partner of childbearing potential, willing to agree to practice a highly effective method of contraception from Visit 2 and at least 3 months after Visit 11 (week 20).
12. Willing to withdraw from any medication for Osteoarthritis including, but not limited to, Opioids, Non-Steroidal Anti-inflammatories (NSAIDs), COX-2 inhibitors, Topical medication, and Duloxetine.
13. Participant agrees to take only the allowed Rescue Medications from the start of the Diary Run-In Period through study completion (maximum 4000 mg paracetamol per day).

Exclusion Criteria:

1. Presence of OA of other major joints (including but not limited to nontarget knee) that could interfere with assessment of pain due to OA of the target knee, in the opinion of the investigator.
2. Current comorbid condition, other than OA, known to be significantly associated with arthritis or joint pathology, including but not necessarily limited to autoimmune disease with significant joint involvement (e.g., Rheumatoid Arthritis or Paget's disease; Seronegative Spondyloarthropathies (e.g. Ankylosing Spondylitis, Psoriasis arthritis, Reactive arthritis); or other systemic disease involving the target knee (including endocrinopathies).
3. The following conditions should be excluded: Known presence of rapidly Progressive Osteoarthritis (RPOA), primary osteonecrosis (including spontaneous osteonecrosis of the knee), subchondral insufficiency fractures (SIF), avascular necrosis, osteoporotic fractures, atrophic OA, excessive malalignment of the knee (anatomical axis angle greater than 10 degrees), pathological fractures, or stress fracture or reaction, vertical tear of the posterior meniscal root, or large or extensive subchondral cysts, or target knee anserine or patellar bursitis of clinical relevance
4. Hip dislocation and congenital hip dysplasia with degenerative joint disease should be excluded.
5. History of gout with recent (< 6 months) pain flares and uncontrolled uric acid levels. Participants with a history or diagnosis of pseudogout (calcium pyrophosphate dihydrate crystal deposition disease) can enroll if there has not been a flare within 6 months prior to screening and use of NSAIDs is not required for management of this condition.
6. Presence of neuropathic pain deemed likely to interfere with trial endpoints, complex regional pain syndrome, or chronic widespread pain syndromes e.g., fibromyalgia.
7. History of significant trauma (e.g., intra-articular fracture) or surgery (excluding injection therapies and arthroscopy) to a knee, hip, or shoulder within the previous 1 year
8. Planned major surgery or other major invasive procedures while participating in the study.
9. Surgery or stent placement for coronary artery disease in the six months prior to screening .
10. Nondiagnostic arthroscopy performed on the target knee joint within 180 days prior to Screening; or diagnostic arthroscopy performed on the target knee joint within 90 days prior to Screening.
11. Intraarticular injection therapies to the target knee joint within 12 weeks prior to Screening, or to any non-target joint within 6 weeks prior to Screening.
12. Participants likely to be deemed unfit for joint replacement surgery due to concomitant illness, in the investigator opinion.
13. Opioid use, including Tramadol, of 4 or more instances per week over the month prior to Screening.
14. Known history of hypersensitivity to monoclonal antibodies.
15. Presence of any medical condition or unstable health status that, in the judgment of the investigator, might adversely impact the safety of the participant.
16. Signs and symptoms of significant cardiac disease, including but not limited to established ischemic heart disease, peripheral arterial disease and /or cerebrovascular disease (unstable angina, myocardial infarction, cardiovascular thrombotic events, transient ischemic attacks, and stroke in the six months prior to screening)
17. Active malignancy or history of malignancy within the past 5 years, with exception of resected and cured basal cell carcinoma and squamous cell carcinoma of the skin.
18. Clinically significant abnormal laboratory parameter(s) and/or ECG parameter(s) during Screening, that, in the judgment of the Investigator, would preclude the participant from participation in this study.
19. Participation in other studies involving investigational drug(s) within 30 days (or 90 days for biologics) prior to screening.
20. History of Carpal Tunnel Syndrome with symptoms within one year of Screening or a Boston Carpal Tunnel Questionnaire (Symptom Severity Scale) mean score ≥3.
21. A total Symptom Impact score on the Survey of Autonomic Symptoms ≥3.
22. Pregnant or breast feeding.
23. Previously received any form of anti-NGF
24. Requires walker or wheelchair for mobility (walking stick permitted).
25. Active or historic substance abuse within one year of Screening in the opinion of the Investigator.
26. Medical history within 5 years of Screening that involves suicidal ideation, suicide attempt, or increased risk of suicide as assessed by the Investigator.
27. Presence of any contraindication to MRI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Westbrook, Study Director — Levicept
Locations (13):
- Czechia (3):
  - CCR Brno, s.r.o, Brno
  - CCR Czech a.s, Pardubice
  - CCR Prague, s.r.o, Prague
- Denmark (3):
  - Sanos Clinic Nordjylland, Gandrup
  - Sanos Clinic Herlev, Herlev
  - Sanos Clinic Syddanmark, Vejle
- Hong Kong Center for Clinical Research, Hong Kong, Hong Kong
- Moldova (2):
  - PMSI Cardiology Institute/RTL SM SRL Consultative ward, Chisinau
  - PMSI Clinical Republican Hospital "Timofei Mosneaga", Chisinau
- Poland (4):
  - NZOZ Bif-Med. s.c., Bytom
  - Somed CR, Lodz
  - Medyczne Centrum Hetmańska, Poznan
  - Somed CR, Warsaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
Started | 130 (1 subject in this group was randomised but intravenous access was not established, therefore the patient never received the study drug. 130 patients are included in efficacy analysis set but only 129 in safety analysis set.) | 130 | 129 | 129
Completed | 120 | 121 | 118 | 116
Not Completed | 10 | 9 | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo | Total
Number analyzed (Participants) | 130 | 130 | 129 | 129 | 518
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 55 | 67 | 46 | 236
  >=65 years | 62 | 75 | 62 | 83 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.68) | 64.5 (8.37) | 63.1 (7.80) | 65.4 (7.8) | 64.0 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 80 | 69 | 76 | 292
  Male | 63 | 50 | 60 | 53 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 12 | 15 | 17 | 22 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 117 | 115 | 112 | 107 | 451
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 12 | 15 | 17 | 22 | 66
  Czechia | 40 | 39 | 30 | 34 | 143
  Denmark | 51 | 50 | 60 | 50 | 211
  Poland | 21 | 24 | 16 | 20 | 81
  Moldova | 6 | 2 | 6 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in WOMAC Pain
Description: The primary efficacy endpoint is the change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score, measured on a 0-10 point scale (0=no pain; 10=worse pain; the result reported is mean change from baseline, therefore the greater the reduction in units the better the outcome)
Time Frame: Week 17 Change from Baseline
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on 0-10 point scale
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
Number analyzed (Participants) | 130 | 130 | 129 | 129
units on 0-10 point scale | -2.77 (0.16) | -2.87 (0.17) | -3.05 (0.17) | -2.26 (0.17)

2. Secondary Outcome: Least Squares Mean Change From Baseline in Post-Staircase Evoked Pain Procedure (StEPP) Pain Intensity
Description: Change from baseline in pain intensity measured following the Staircase Evoked Pain Procedure (StEPP), using a numeric rating scale ranging from 0 to 10 (0=no pain; 10=worse pain; the result reported is mean change from baseline, therefore the greater the reduction in units the better the outcome)
Time Frame: Week 17 Change from Baseline
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on 0-10 pain scale
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
Number analyzed (Participants) | 111 | 119 | 113 | 110
units on 0-10 pain scale | -2.5 (0.20) | -2.6 (0.19) | -3.0 (0.20) | -1.8 (0.20)

3. Secondary Outcome: Least Squares Mean Change From Baseline in WOMAC Physical Function
Description: Change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function subscale, measured on a 0 to 10 point scale (0=no impact on physical function; 10=worse impact on physical function; the result reported is mean change from baseline, therefore the greater the reduction in units the better the outcome)
Time Frame: Week 17 Change from Baseline
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on 0-10 point scale
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
Number analyzed (Participants) | 118 | 119 | 116 | 113
units on 0-10 point scale | -2.40 (0.159) | -2.49 (0.159) | -2.75 (0.162) | -1.84 (0.164)

4. Secondary Outcome: Least Squares Mean Change From Baseline in WOMAC Joint Stiffness Subscale
Description: Change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Joint Stiffness Subscale, scored on a 0 to 10 point scale (0=no stiffness; 10=worst stiffness; the result reported is mean change from baseline, therefore the greater the reduction in units the better the outcome)
Time Frame: Week 17 Change from Baseline
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on 0-10 point scale
Groups:
- Placebo: Intravenous infusion fo saline vehicle as placebo
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
Number analyzed (Participants) | 118 | 119 | 116 | 113
units on 0-10 point scale | -2.60 (0.179) | -2.82 (0.179) | -3.20 (0.182) | -1.75 (0.185)

5. Secondary Outcome: Least Squares Mean Change From Baseline in Patient Global Assessment
Description: Change from baseline in the Patient Global Assessment, measured on a 0 to 10 numeric rating scale where 0 indicates "Very good" and 10 indicates "Very bad". The result reported is the mean change from baseline; therefore, the greater the reduction in units, the better the outcome.
Time Frame: Week 17 Change from Baseline
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on 0-10 point scale
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
Number analyzed (Participants) | 118 | 119 | 116 | 113
units on 0-10 point scale | -2.3 (0.18) | -2.6 (0.18) | -2.8 (0.19) | -1.7 (0.19)

ADVERSE EVENTS:
Time Frame: The AE reporting period for safety surveillance begins when the participant is initially included in the trial (date of signature of ICF) and continues until Week 30
Description: All AEs reported by participants or observed by study personnel from the time of signing the Informed Consent Form through week 30 were documented. Each AE was evaluated for severity using the Qualitative Toxicity Scale, which categorised events as mild, moderate, or severe based on the level of discomfort and impact on the participant's daily activities. Investigators also assessed the relationship between AEs and the IMP, determining whether the event was unrelated or related to the IMP.
Arm/Group | 0.3 mg/kg LEVI-04 | 1.0 mg/kg LEVI-04 | 2.0 mg/kg LEVI-04 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/130 | 0/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129 | 1/130 | 3/129 | 3/129
Other Adverse Events (participants affected / at risk) | 36/129 | 44/130 | 58/129 | 62/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg/kg LEVI-04 (N=129) | 1.0 mg/kg LEVI-04 (N=130) | 2.0 mg/kg LEVI-04 (N=129) | Placebo (N=129)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 | 0
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg/kg LEVI-04 (N=129) | 1.0 mg/kg LEVI-04 (N=130) | 2.0 mg/kg LEVI-04 (N=129) | Placebo (N=129)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 15 | 15 | 20
Nasopharyngitis (Infections and infestations) | 6 | 8 | 13 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 8 | 3
Headache (Nervous system disorders) | 4 | 3 | 8 | 6
Covid-19 (Infections and infestations) | 5 | 2 | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 5 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT05618782/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT05618782/SAP_001.pdf